CLINICAL TRIAL: NCT03962036
Title: Effect of One-lung Ventilation on BIS Values
Status: Terminated | Type: Observational
Why Stopped: Study showed no results
Sponsor: Christopher McKee (Other)
Responsible Party: Sponsor-Investigator, Christopher McKee, Attending Anesthesiologist, Nationwide Children's Hospital
Organization: Nationwide Children's Hospital (Other)
Other Study IDs: STUDY00000324
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Surgery; Thoracic
MeSH Terms: interventions — Consciousness Monitors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Bispectral index monitor — BIS monitor is a novel measure of the level of consciousness by algorithmic analysis of a patient's electroencephalogram during general anesthesia.
  Other Names: BIS

SUMMARY:
In this observational study, all enrolled patients having a thoracic surgical procedure requiring lung isolation will have a bispectral index (BIS) monitor placed at time of induction. BIS monitors are used to assist in determining depth of anesthesia. This study will evaluate changes in BIS before, during and after lung isolation.

ELIGIBILITY:
Inclusion Criteria:

* Patients coming for thoracic surgery with anticipated need for lung isolation

Exclusion Criteria:

* None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Surgical patients requiring one lung ventilation at Nationwide Children's Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2019-10-11 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Change in BIS | From baseline to one lung ventilation (average time frame of 30 mins. - 1 hr.)
  Comparing the BIS readings while on two lung ventilation to the BIS readings after switching the one lung ventilation.

CONTACTS AND LOCATIONS:
Locations (1):
- Nationwide Children's Hospital, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No